CLINICAL TRIAL: NCT03167476
Title: Comparative Study of microRNA Changes in Patients With Reactive Lymphoid Hyperplasia and Malignant Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Collaborators: Chengdu Nuoen Biotechnologies, Inc. (Other); Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Uestc502
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2016-08

CONDITIONS: Lymphoma; Hyperplasia Lymphoid Reactive
Keywords: miRNA; biomarker
MeSH Terms: conditions — Lymphoma; Pseudolymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RLH: This group includes subjects diagnosed with reactive lymphoid hyperplasia.
- Lymphoma: This group includes subjects diagnosed with lymphoma.

SUMMARY:
The objectives are to:

1. validate a panel of tissue-specific miRNAs that are differentially expressed in the tissue of patients with and without reactive hyperplasia and lymphoma.
2. investigate the physiological range of the miRNA panel in lymphoma and reactive hyperplasia subjects.
3. investigate the dysregulation of miRNA panel and their prognostic and predictive values in clinical outcomes to identifying patients with malignant lymphoma or reactive hyperplasia.

The objectives are to:

1. validate a panel of tissue-specific miRNAs that are differentially expressed in the tissue of patients with and without reactive hyperplasia and lymphoma.
2. investigate the physiological range of the miRNA panel in lymphoma and reactive hyperplasia subjects.
3. investigate the dysregulation of miRNA panel and their prognostic and predictive values in clinical outcomes to identifying patients with malignant lymphoma or reactive hyperplasia.

This trial involves tissue samples diagnosed as lymphoma and reactive hyperplasia. The investigators will develop panels of miRNAs that are specific biomarkers of lymphoma, and assist clinical outcomes with these miRNAs.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and above
* Has condition related to lymphoma or reactive lymphoid hyperplasia

Exclusion Criteria:

* Age below 18 years
* Known pregnancy
* lymph tissue cannot be accessed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research project will recruit a cohort of observational lymphoma patients. Diagnosis and immunophenotyping should be performed on FFPE tissues according to the WHO-classification system and reviewed by an in-house pathologist. Reactive hyperplasia controls will also be recruited to demonstrate the physiological level of different body-tissue miRNAs.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
The concentration of miRNA expression quantitated in absolute copy numbers and their correlation in patients with reactive hyperplasia and lymphoma. | Three years
  The concentration of tissue miRNAs in absolute quantification in comparison to reactive hyperplasia and lymphoma. To investigate the potential prognosis of lymphoma by the expression difference of the miRNA panel. Sensitivity, specificity and the potential scopes of selected miRNA in the miRNA panel to distinguish hyperplasia and lymphoma and against standard clinical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, PhD, Study Director — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China